CLINICAL TRIAL: NCT02238743
Title: A Single-Arm, Case-Series to Determine the Feasibility of Safe Skills Transfer for Laparoscopic Ventral Hernia Repair Utilizing a Hands-On Proctorship Model.
Brief Title: Assuring and Defining Outcomes Through Procedural Training Using a Proctorship Model That Collects Patient Outcomes A Single-Arm, Case-Series to Determine the Feasibility of Safe Skills Transfer for Laparoscopic Ventral Hernia Repair Utilizing a Hands-On Proctorship Model.
Acronym: ADOPT
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: Project ADOPT- UM
Record Dates: First submitted 2014-08-21; First posted 2014-09-12 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the Project ADOPT- Ventral Hernia case-series is to collect clinical outcome data following the completion of a hands-on proctorship training model in laparoscopic ventral hernia repair.

DETAILED DESCRIPTION:
The ADOPT- Ventral Hernia project is designed as a prospective, single arm, case series. The proctor will select a limited number of licensed surgeon trainees (up to 5) as agreed upon by Covidien and the proctor. The proctor will then train through clinical immersions, hands on proctorship and video training for proper technique on minimally invasive surgical (MIS) repair of ventral hernia. After the training, the data will be collected on the trainee's next 10 MIS ventral hernia repair cases, pending subject consent to collect data. Procedural and Post-Operative details will be captured for each of these subjects who have undergone the laparoscopic ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Determined by surgeon's standard of care

Exclusion Criteria:

* Determined by surgeon's standard of care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Determined by surgeon
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of complications during independent cases post proctorship | up to 30 days
  collect clinical outcome data following the completion of a hands-on proctorship training model in laparoscopic ventral hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Pearl, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States